CLINICAL TRIAL: NCT05395390
Title: Circuit-Exercise Training on Subjects With and Without Chronic Respiratory Disease
Brief Title: COPD Circuit Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Responsible Party: Principal Investigator, Marielle PKJ Engelen, PhD, Professor, Texas A&M University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-0149
Record Dates: First submitted 2021-12-10; First posted 2022-05-27 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: OSA; Covid19; Residual Symptoms of COVID 19; COPD
MeSH Terms: conditions — COVID-19; Pulmonary Disease, Chronic Obstructive | interventions — Exercise; Resistance Training

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Exercise (Resistance Training — Resistance Training done both at home and on site using either dumbells or keiser pneumatic exercise machines respectively

SUMMARY:
This study is being done to understand body's response to hybrid home-based and on-site rehabilitation program utilizing individually tailored exercises throughout a total of 18 sessions with 12 of them occurring onsite, in people with and without chronic respiratory diseases, such as Chronic Obstructive Pulmonary Disease (COPD) and Obstructive Sleep Apnea (OSA) and in individuals recovered from COVID-19. Exercise training programs vary widely for people with COPD, OSA, and during prolonged recovery from COVID infection. This study will help identify if this program is helpful to address muscle loss and fatigue specifically in populations with and without chronic respiratory diseases.

ELIGIBILITY:
Inclusion Criteria:

* Ability to walk, sit down and stand up independently

  * Age 30 - 85 years
  * Ability to lay in supine or elevated position for up to 3 hours
  * Diagnosis of moderate to very severe chronic airflow limitation and compliant to the following criteria: FEV1 < 70% of reference FEV1

-or- Obstructive Sleep Apnea (OSA)

-or- 2 weeks post-recovered* from laboratory confirmed case of COVID

● Willingness and ability to comply with the protocol

*Recovered is defined according to Brazos County Health District as someone who has been fever-free for 24 hours without fever-reducing medications, and it has been 10 days after onset of symptoms.

Inclusion criteria control subjects

* Healthy male or female according to the investigator's or appointed staff's judgment
* Ability to walk, sit down and stand up independently
* Age 30 - 85 years
* Ability to lay in supine or elevated position for up to 3 hours
* No diagnosis of chronic lung disease
* Willingness and ability to comply with the protocol

Exclusion Criteria:

* Unable to exercise due to physical limitations (i.e. neuromuscular and/or orthopedic disorders)

  * Established diagnosis of malignancy
  * Presence of acute illness or metabolically unstable chronic illness
  * Presence of fever within the last 3 days.
  * Expected to have surgery within 1 month of screening or during exercise training
  * Any other condition according to the PI or research staff that was found during the screening visit, that would interfere with the study or safety of the patient.
  * Previous injury that could interfere with participation in resistance exercise protocol.
  * Failure to give informed consent or Investigator's uncertainty about the willingness or ability of the subject to comply with the protocol requirements.
  * (Possible) pregnancy.
  * Already enrolled in another clinical trial and that clinical trial interferes with participating in this study. When during the period from enrollment to the test day any condition causing the subject to not meet inclusion criteria or to meet exclusion criteria, the subject will be excluded from the study.

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2021-02-02 (Actual); Primary Completion 2023-08-07 (Actual); Study Completion 2023-08-07 (Actual)

PRIMARY OUTCOMES:
Whole-body protein and amino acid metabolism response to training | up to 8 weeks Exercise Intervention
  Whole-body production rate measured after stable tracer administration

SECONDARY OUTCOMES:
Body Composition using Dual Energy X-Ray Absorptiometry bone density | up to 8 week Exercise Intervention
  Measurement of bone mineral density (g/cm^2)between COPD patients and healthy older adults using DXA
Body Composition using Dual Energy X-Ray Absorptiometry Muscle | up to 8 week Exercise Intervention
  Measurement of muscle mass (kg)
Body Composition using Dual Energy X-Ray Absorptiometry Fat | up to 8 week Exercise Intervention
  Measurement of fat mass (kg)
Bone mineral density by BIA | up to 8 week Exercise Intervention
  Differences in muscle mass (kg), fat mass (kg), and extra- and intracellular fluid (L) between COPD patients and healthy older adults using BIA.
Handgrip strength dynamometry by Handgrip Dynamometer | up to 8 week Exercise Intervention
  Difference and changes in handgrip strength pre and post exercise
6 minute walk test distance by 6 minute walk test | up to 8 week Exercise Intervention
  With this sub-maximal exercise test, aerobic capacity and endurance will be compared between COPD patients and healthy older adults. The outcome is the distance covered over a time of 6 minutes.
Skeletal muscle strength of leg by Kin-Com | up to 8 week Exercise Intervention
  Difference in muscle strength of leg using kin-com machine between pre and post exercise intervention.
C-reactive protein by Blood Analysis | up to 8 week Exercise Intervention
  Differences and changes in the concentration of the inflammatory marker C-reactive protein
Attention and executive functions measured by Trail Making Test (TMT) | up to 8 week Exercise Intervention
  In Part A, the examinee is instructed to connect a set of 25 circles with numbers as quickly as possible while maintaining accuracy. In Part B, the examinee is instructed to connect a set of 25 circles, alternating between numbers and letters, as quickly as possible while maintaining accuracy. Measures attentional resources and is a measure of the frontal lobe "executive" functions of visual search, set-switching and mental flexibility. The total time in seconds will be recorded for each measure.
Attention and executive functions measured by Stroop Color-Word Test (SCWT) | up to 8 week Exercise Intervention
  A word page with words printed in black ink, a color page with blocks printed in color, and a color-word page where the color and the word do not match. The examinee reads the words or names the ink colors as quickly as possible within a time limit. Measures selective attention and inhibitory control. The total time in seconds was reported for each trial.
Gut function as reported by "The Gastrointestinal Symptom Rating Scale" | up to 8 week Exercise Intervention
  Self-administered questionnaire regarding gut function and associated symptoms. It is composed of 15 items (7-Point Likert Scale) assessing Reflux, Abdominal pain, Indigestion, Diarrhoea and Constipation. Scores range from 15 to 105 with a higher score indicating more discomfort.
Physical activity as reported by "Physical Activity Scale for the Elderly | up to 8 week Exercise Intervention
  Self-administered questionnaire is intended for use in an elderly population and focuses on 3 types of activities: leisure time activities, household activities and work-related activities.
State of mood as measured by the Hospital Anxiety and Depression Scale (HADS) | up to 8 week Exercise Intervention
  A fourteen item self-assessment scale. Seven of the items related to anxiety and seven relate to depression. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 (no symptoms) and 21 (severe symptoms) for either anxiety or depression.
COPD Assessment Test | up to 8 week Exercise Intervention
  Self-administered questionnaire regarding impact of COPD on daily life
3-day diet diary | up to 8 week Exercise Intervention
  The subject is asked to note in detail all the food and drinks consumed during 3 days (2 week days and 1 weekend day) in the week prior to each test day.
Group differences in learning and memory as measured by Digit Span | up to 8 week Exercise Intervention
  Recall of numbers in the same order (Digit Forward) and in reverse order (Digit Backward). Measures auditory attention and verbal working memory.
Group differences in overall cognitive abilities as measured by Montreal Cognitive Assessment (MoCA) | up to 8 week Exercise Intervention
  Assesses several cognitive domains and is used for the screening of mild cognitive impairment. Total scores range from 0-30 with lower scores indicating decreased functioning.
Group differences in state of mood as measured by the Profile of Mood State (POMS) | up to 8 week Exercise Intervention
  A psychological distress scale to measure mood disturbance in 6 domains - fatigue-inertia, vigor-activity, tension-anxiety, depression-dejection, anger-hostility, and confusion-bewilderment.
Group differences in learning and memory as measured by Controlled Oral Word Association Test (COWAT) | up to 8 week Exercise Intervention
  The examinee is required to say as many words as they can think of in one minute that begin with a given letter of the alphabet. The task contains three trials. Measures phonemic verbal fluency. The raw score (total and mean words recorded across the three trials) will be reported.
Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) | up to 8 week Exercise Intervention
  Quality of life concerns related to fatigue will be assessed only in COPD patients with this questionnaire.
Peak Power and Strength by Keiser Resistance Training Equipment | up to 8 week Exercise Intervention
  Changes in Peak Power and Strength measured through testing completed using Keiser Pneumatic Resistance Training Devices

CONTACTS AND LOCATIONS:
Locations (1):
- Texas A&M University, College Station, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
Data may be shared upon request for up to 6 years beyond completion of the trial based on methods/proposal approved by both parties' institutional review committees. Individual participant data that underlie the results of the trial may be shared after de-identification (text, tables, figures, and appendices). Additional documents available per request include: study protocol, statistical analysis plan, and informed consent. Requests should be directed to Dr. Marielle Engelen (mpkj.engelen@ctral.org).

REFERENCES:
- [Derived] Yu AK, Deutz NEP, Perez CN, DeWandel S, Ruebush LE, Engelen MPKJ. The acute effects of alpha-lactalbumin intake on tryptophan metabolites and mood in older adults with Mild Cognitive Impairment. Nutr Neurosci. 2025 Sep 14:1-15. doi: 10.1080/1028415X.2025.2554359. Online ahead of print. PMID 40946231